CLINICAL TRIAL: NCT07075575
Title: Smoking Cessation Among Native Hawaiians: A Test of Pharmacotherapies and Group-Based Counseling
Brief Title: Quit-Smoking Study for Native Hawaiians
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POKHREL-2024-1
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Tobacco Use Disorder; Smoking Cessation
Keywords: Native Hawaiian; Smoking cessation; Nicotine replacement therapy; Nicotine gum; Cigarette Smoking; Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NRT Gum Only (Experimental): Participants receive nicotine gum (2 mg) according to a 12-week FDA-approved tapering schedule. No counseling is provided.
  Interventions: Drug: Nicotine Polacrilex Gum (2 mg)
- CBGT Only (Experimental): Participants attend six weekly sessions of cognitive-behavioral group therapy (CBGT) for smoking cessation. No nicotine gum is provided.
  Interventions: Behavioral: Cognitive Behavioral Group Therapy (CBGT)
- CBGT + NRT Gum (Experimental): Participants receive both nicotine gum (2 mg, tapered over 12 weeks) and attend six weekly CBGT sessions for smoking cessation.
  Interventions: Drug: Nicotine Polacrilex Gum (2 mg); Behavioral: Cognitive Behavioral Group Therapy (CBGT)

INTERVENTIONS:
Drug: Nicotine Polacrilex Gum (2 mg) — Participants chew 2 mg nicotine gum according to a tapering 12-week schedule: Weeks 1-6: 1 piece every 1-2 hours; at least 9 pieces/day; Weeks 7-9: 1 piece every 2-4 hours; Weeks 10-12: 1 piece every 4-8 hours. Max 24 pieces/day. Gum is distributed every 2 weeks during study visits.
  Arm(s) Used In:
  NRT Gum Only CBGT + NRT Gum
  Arms: CBGT + NRT Gum; NRT Gum Only
Behavioral: Cognitive Behavioral Group Therapy (CBGT) — Participants attend six sessions of group-based cognitive behavioral therapy focused on smoking cessation, over the 12-week study period. Sessions include education on cravings, relapse prevention, stress management, and self-efficacy building.
  Arm(s) Used In:
  CBGT Only CBGT + NRT Gum
  Arms: CBGT + NRT Gum; CBGT Only

SUMMARY:
This study aims to help Native Hawaiian adults quit smoking by testing two common methods: nicotine gum and group-based counseling. Participants will be assigned to one of three groups: (1) nicotine gum only, (2) group counseling only, or (3) a combination of both. The study will take place at public housing sites on O'ahu. Researchers will check if these approaches-alone or in combination-can support people in successfully quitting smoking. The goal is to find out which method works best and is most acceptable in this community.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as full or part Native Hawaiian
* Between the ages of 18 and 80 years, inclusive, at eligibility screening
* Currently smoking ≥5 cigarettes per day (self-report) at eligibility screening
* Has smoked more than 100 cigarettes in his/her lifetime (self-report)
* Affiliated with one of three (3) designated public housing complexes at which the intervention will be delivered: Kalihi Valley Homes, Kuhio Park Terrace, Mayor Wright Housing
* Willing to make a smoking cessation attempt the day after the first study visit (i.e., date of consent)
* Willing to engage in use of nicotine replacement therapy gum (NRT gum) and/or smoking cessation-focused cognitive-behavioral group therapy (CBGT)
* Participant must agree to not use any form of pharmacotherapy (i.e., prescription medication or any form of nicotine replacement therapy) to try to quit smoking during the 12-week study period, except as specifically assigned to his or her study condition and distributed by the research team
* Participant must agree to not use other tobacco or nicotine products (e.g., cigars, little cigars, electronic cigarettes, nicotine pouches) during the 12-week study period
* Participant must agree to not smoke or vape cannabis (i.e., marijuana) during the 12- week study period
* Participant must agree to not use other illicit drugs, including prescription opioid medications, during the 12-week study period
* Participant must be able to speak, read, and write English
* Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent

Exclusion Criteria:

* Pregnant or nursing, or planning to become pregnant or breastfeed in the next three (3) months
* Use of pharmacotherapy (i.e., prescription medication or any form of nicotine replacement therapy) to try to quit smoking in the 30 days prior to eligibility screening
* Use of other tobacco or nicotine products (e.g., cigars, little cigars, electronic cigarettes, nicotine pouches) in the 30 days prior to eligibility screening
* Use of smoked or vaped cannabis (i.e., marijuana) in the 30 days prior to eligibility screening
* Use of other illicit drugs, including prescription opioid medications, in the 30 days prior to eligibility screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence abstinence (PPA) | 12 weeks after baseline (Study Visit 8)
  Self-reported 7-day point prevalence abstinence from cigarette smoking, confirmed by exhaled carbon monoxide (eCO) <10 ppm at final follow-up visit.

SECONDARY OUTCOMES:
Change in nicotine dependence | Baseline to 12 weeks
  Change in nicotine dependence scores as measured by standardized tools (e.g., Fagerström Test for Nicotine Dependence).
Change in smoking self-efficacy | Baseline to 12 weeks
  Change in participants' confidence in their ability to quit smoking, measured using a validated smoking self-efficacy scale.
Number of adverse events | Throughout the 12-week intervention period
  Frequency and severity of adverse events related to nicotine gum or study procedures, as reported by participants or observed by study staff.

CONTACTS AND LOCATIONS:
Overall Officials: Crissy T Kawamoto, Study Director — University of Hawai'i Cancer Center; Pallav Pokhrel, PhD, MPH, Principal Investigator — University of Hawai'i Cancer Center
Locations (1):
- University of Hawai'i, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Result] Webb MS, de Ybarra DR, Baker EA, Reis IM, Carey MP. Cognitive-behavioral therapy to promote smoking cessation among African American smokers: a randomized clinical trial. J Consult Clin Psychol. 2010 Feb;78(1):24-33. doi: 10.1037/a0017669. PMID 20099947
- [Result] Stead LF, Carroll AJ, Lancaster T. Group behaviour therapy programmes for smoking cessation. Cochrane Database Syst Rev. 2017 Mar 31;3(3):CD001007. doi: 10.1002/14651858.CD001007.pub3. PMID 28361497
- [Result] Rohsenow DJ, Martin RA, Tidey JW, Colby SM, Monti PM. Treating Smokers in Substance Treatment With Contingent Vouchers, Nicotine Replacement and Brief Advice Adapted for Sobriety Settings. J Subst Abuse Treat. 2017 Jan;72:72-79. doi: 10.1016/j.jsat.2016.08.012. Epub 2016 Aug 18. PMID 27658756
- [Result] Ong JC, Kuo TF, Manber R. Who is at risk for dropout from group cognitive-behavior therapy for insomnia? J Psychosom Res. 2008 Apr;64(4):419-25. doi: 10.1016/j.jpsychores.2007.10.009. PMID 18374742
- [Result] Nevid JS, Javier RA. Preliminary investigation of a culturally specific smoking cessation intervention for Hispanic smokers. Am J Health Promot. 1997 Jan-Feb;11(3):198-207. doi: 10.4278/0890-1171-11.3.198. PMID 10165099
- [Result] Meredith SE, Grabinski MJ, Dallery J. Internet-based group contingency management to promote abstinence from cigarette smoking: a feasibility study. Drug Alcohol Depend. 2011 Oct 1;118(1):23-30. doi: 10.1016/j.drugalcdep.2011.02.012. Epub 2011 Mar 16. PMID 21414733
- [Result] Lo Coco G, Melchiori F, Oieni V, Infurna MR, Strauss B, Schwartze D, Rosendahl J, Gullo S. Group treatment for substance use disorder in adults: A systematic review and meta-analysis of randomized-controlled trials. J Subst Abuse Treat. 2019 Apr;99:104-116. doi: 10.1016/j.jsat.2019.01.016. Epub 2019 Jan 24. PMID 30797382
- [Result] Lee PN, Fariss MW. A systematic review of possible serious adverse health effects of nicotine replacement therapy. Arch Toxicol. 2017 Apr;91(4):1565-1594. doi: 10.1007/s00204-016-1856-y. Epub 2016 Oct 3. PMID 27699443
- [Result] Lancaster T, Stead LF. Individual behavioural counselling for smoking cessation. Cochrane Database Syst Rev. 2017 Mar 31;3(3):CD001292. doi: 10.1002/14651858.CD001292.pub3. PMID 28361496
- [Result] Hunt DF, Bailey J, Lennox BR, Crofts M, Vincent C. Enhancing psychological safety in mental health services. Int J Ment Health Syst. 2021 Apr 14;15(1):33. doi: 10.1186/s13033-021-00439-1. PMID 33853658
- [Result] Hiscock R, Murray S, Brose LS, McEwen A, Bee JL, Dobbie F, Bauld L. Behavioural therapy for smoking cessation: the effectiveness of different intervention types for disadvantaged and affluent smokers. Addict Behav. 2013 Nov;38(11):2787-96. doi: 10.1016/j.addbeh.2013.07.010. Epub 2013 Jul 21. PMID 23954946
- [Result] Goldstein AO, Gans SP, Ripley-Moffitt C, Kotsen C, Bars M. Use of Expired Air Carbon Monoxide Testing in Clinical Tobacco Treatment Settings. Chest. 2018 Feb;153(2):554-562. doi: 10.1016/j.chest.2017.11.002. Epub 2017 Nov 11. PMID 29137909
- [Result] Gifford EV, Kohlenberg BS, Hayes SC, Pierson HM, Piasecki MP, Antonuccio DO, Palm KM. Does acceptance and relationship focused behavior therapy contribute to bupropion outcomes? A randomized controlled trial of functional analytic psychotherapy and acceptance and commitment therapy for smoking cessation. Behav Ther. 2011 Dec;42(4):700-15. doi: 10.1016/j.beth.2011.03.002. Epub 2011 May 25. PMID 22035998
- [Result] Creamer MR, Wang TW, Babb S, Cullen KA, Day H, Willis G, Jamal A, Neff L. Tobacco Product Use and Cessation Indicators Among Adults - United States, 2018. MMWR Morb Mortal Wkly Rep. 2019 Nov 15;68(45):1013-1019. doi: 10.15585/mmwr.mm6845a2. PMID 31725711
- [Result] Carter RE, Sonne SC, Brady KT. Practical considerations for estimating clinical trial accrual periods: application to a multi-center effectiveness study. BMC Med Res Methodol. 2005 Mar 30;5:11. doi: 10.1186/1471-2288-5-11. PMID 15796782
- [Result] Babb S, Malarcher A, Schauer G, Asman K, Jamal A. Quitting Smoking Among Adults - United States, 2000-2015. MMWR Morb Mortal Wkly Rep. 2017 Jan 6;65(52):1457-1464. doi: 10.15585/mmwr.mm6552a1. PMID 28056007
- See also: General consumer information about nicotine gum, including proper use, precautions, and side effects. Provided by MedlinePlus, a service of the U.S. National Library of Medicine. — https://medlineplus.gov/druginfo/meds/a684056.html
- See also: Strategic plan from the Hawai'i State Department of Health outlining goals and priorities for tobacco prevention and control across the state, including culturally tailored interventions for Native Hawaiians and other priority populations. — https://hhsp.hawaii.gov/assets/pdf/HHSP_Tobacco_Plan_WEB.pdf
- See also: Behavioral Risk Factor Surveillance System (BRFSS) data from the Hawai'i Health Data Warehouse showing smoking prevalence among adults by race/ethnicity from 2018-2023. Useful for understanding disparities in tobacco use among Native Hawaiians and other — https://hhdw.org/report/query/result/brfss/SmokeCurrent/SmokeCurrentCrude11_.html
- See also: Summary report from the Hawai'i Tumor Registry presenting cancer incidence and mortality data in Hawai'i from 2014-2018. Includes statistics by race/ethnicity and geographic region, supporting local relevance of tobacco-related cancer prevention. — https://uhcancercenter.org/pdf/htr/Cancer%20at%20a%20Glance%202014-2018.pdf
- See also: ICH E2A guideline outlining international standards for defining, collecting, and reporting clinical safety data, including serious adverse events (SAEs) and expedited reporting procedures. — https://database.ich.org/sites/default/files/E2A_Guideline.pdf
- See also: Guidelines from the National Cancer Institute (NCI) detailing adverse event reporting requirements for investigators conducting studies under NCI's Division of Cancer Treatment and Diagnosis (DCTD) and Division of Cancer Prevention (DCP) INDs and IDEs. — https://ctep.cancer.gov/protocolDevelopment/electronic_applications/docs/aeguidelines.pdf
- See also: Official NCI Thesaurus entry for "Nicotine Dependence," providing standardized terminology and coding used in biomedical research and clinical trial reporting. — https://ncit.nci.nih.gov/ncitbrowser/ConceptReport.jsp?dictionary=NCI_Thesaurus&ns=NCI_Thesaurus&code=C41331#
- See also: National Cancer Institute fact sheet offering practical guidance for managing nicotine withdrawal symptoms and behavioral triggers when quitting tobacco. Intended for patients and healthcare providers. — https://www.cancer.gov/about-cancer/causes-prevention/risk/tobacco/withdrawal-fact-sheet#r1
- See also: The 2014 Surgeon General's Report summarizes 50 years of scientific evidence on the health effects of smoking. It provides comprehensive data on smoking-related diseases, tobacco use patterns, and public health impact in the U.S. — https://www.ncbi.nlm.nih.gov/books/NBK179276/pdf/Bookshelf_NBK179276.pdf